CLINICAL TRIAL: NCT07230496
Title: A Phase I, Randomized, Double-blind, Placebo-Controlled Study Evaluating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of LAE103 as Single and Multiple Ascending Doses in Healthy Overweight/Obese Participants, and as Single Dose in Healthy Postmenopausal Women, With an Additional Evaluation of Single Ascending Dose of LAE103 in Combination With LAE102 in Healthy Overweight/Obese Participants
Brief Title: A Study to Investigate Safety, Tolerability and Pharmacokinetics of LAE103 or LAE103 in Combination With LAE102 in Healthy Overweight/Obese Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Laekna Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: LAE103INT1001
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment arm of single drug (Experimental): LAE103 injection, subcutaneous (SC) injection
  Interventions: Drug: LAE103 injection; Drug: Saline
- comparator arm (Placebo Comparator): Saline
  Interventions: Drug: Saline
- Treatment arm of combination (Experimental): LAE102 injection combined with LAE103 injection, single dose, subcutaneous (SC) injection
  Interventions: Drug: LAE102 injection in combined with LAE103 injection; Drug: Saline

INTERVENTIONS:
Drug: LAE103 injection — subcutaneous injection of LAE103 alone
  Arms: Treatment arm of single drug
Drug: LAE102 injection in combined with LAE103 injection — LAE102 injection in combined with LAE103 injection via subcutaneous
  Arms: Treatment arm of combination
Drug: Saline — Saline via subcutaneous

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of LAE103 injection in healthy overweight/obese participants or healthy postmenopausal women. Study will also evaluate the safety, tolerability and preliminary pharmacodynamic effect of multiple dose injections in overweight/obese participants.

In addition, the study will also investigate the safety, tolerability of a single-dose co-administration of LAE102 and LAE103 in healthy overweight/obese participants.

DETAILED DESCRIPTION:
This is a randomized, double-blind study comprising of a single-dose escalation study in healthy overweight/obese participants (Part A), a single dose study in healthy postmenopausal women (Part B), and a multiple-dose escalation study in healthy overweight/obese participants (Part C), designed to evaluate the safety, tolerability, Pharmacokinetics (PK )and pharmacodynamics (PD) profiles of LAE103 administered alone.

In addition, the study will also investigate the safety, tolerability, and PK/PD profiles of a single-dose co-administration of LAE102 and LAE103 in healthy overweight/obese participants (Part D).

About 104 participants will be enrolled in 13 cohorts with each cohort including 8 participants randomized 6:2 study drug:Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Are capable of giving signed informed consent and comply with the requirements and restrictions listed in the ICF and in this protocol.
* Male or female participants aged 18 to 55 years in part A, C, D. Female participants aged 45 to 75 years in Part B.
* Have a BMI within the range of 25.0 to 40.0 kg/m2 in Parts A, C, and D and a BMI within the range of 20.0 to 35.0 kg/m2 in Part B.
* Participants without childbearing potential or Participants with childbearing potential, non-pregnant, non-lactating, must agree to use two forms of effective methods of contraception (at least one form must be highly effective) .
* Male participants with female partners of childbearing potential must agree to use adequate methods of contraception. Male subjects are not allowed to donate sperm during this trial.
* Are overtly healthy participants or Have FSH levels ≥ 40 IU/L at screening (Part B only).
* Are willing to make themselves available for study visits for the duration of the study and are willing to follow study procedures.

Exclusion Criteria:

* Have a history or presence of clinically significant medical condition(s).
* Have a history of any malignancy within the past 5 years. other than basal cell or squamous epithelial carcinomas in situ and cervical carcinoma in situ that have been resected with no evidence of metastatic diseases for 3 years.
* Have a fasting serum triglyceride level of more than 500 mg/dL(5.6 mmol/L) at screening.
* Estimated glomerular filtration rate (eGFR) less than 90 mL/min/1.73 m2 at screening for Part A, C, and Part D or less than 60 mL/min/1.73 m2 at screening for Part B.
* Have an abnormality in the 12-lead ECG to increase risk or QT (QTcF) interval greater than 450 msec at screening.
* Have an abnormal blood pressure.
* Positive human HIV antibodies or positive hepatitis C antibodies or positive hepatitis B surface antigen.
* A history of, or known hypersensitivity to antibody drug, study procedure or any severe food or drug allergies.
* Underwent major surgery within 30 days prior to study intervention administration or plan to undergo major surgery during the study.
* Self-reported weight change is more than 5% in the previous 3 months prior to screening.
* Engaged in regular weightlifting, fitness, or strength training aimed at enhancing muscle strength.
* Use of GLP-1 receptor agonists, or weight loss medication within 3 months prior to the first dose of the investigational product.
* Have used in the past 90 days (before screening) or intend to use during the study any medication that may affect FSH levels.
* Have used or intend to use prescription or over the counter medications, or herbal medicines, from 14 days or 5 half-lives (if known), whichever is longer, prior to study intervention administration until the last visit.
* Received any vaccine 30 days prior to screening or plan to receive any vaccine during the study.
* Have participated, are currently enrolled in, or discontinued from a clinical trial involving an investigational drug or device or off-label use of a drug or device within the last 90 days, or 5-half-lives (if known, whichever is longer), of the last administration of study drug or application of the device, or any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have previously completed or withdrawn from this study or any other study investigating this study intervention.
* Have an average weekly alcohol consumption exceeding 14 units per week for female participants, 21 units per week for male participants, or positive alcohol test at screening or admission, or a history of alcohol abuse disorder within 1 year prior to screening, or an inability or unwillingness to stop alcohol consumption 7 days prior to dosing.
* Have known or suspected history of substance abuse or test positive for drugs of abuse at screening or admission.
* Are smoking more than 5 cigarettes (or the equivalent of other tobacco products) per day within 90 days prior to screening, or unable or unwilling to stop smoking tobacco products during the confinement period.
* Have donated blood or experienced blood loss of more than 400 mL within 30 days prior to screening.
* Are fasting or receiving weight loss treatment within 30 days prior to study intervention administration, or experiencing major changes in lifestyle.
* In the opinion of the investigator or Sponsor and medical monitor, are unsuitable for inclusion in the study.
* Are Laekna Limited. employees, CRO employees, investigator, or site personnel directly affiliated with this study or the immediate families of any of these. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
* Have contraindications for MRI scan or do not meet the requirements for MRI scan as per local guideline. (This criterion applies only to Parts C and D.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 104 (Estimated)
Dates: Start 2025-12-30 (Actual); Primary Completion 2028-03-20 (Estimated); Study Completion 2028-03-20 (Estimated)

PRIMARY OUTCOMES:
Number & severity of participants with treatment-related adverse events | From Day1 to Day70 for single dose part. From Day 1 to Day98 for multiple dose part
  Findings on physical examination, ECG, vital signs, and reports of the laboratory results via investigator assessment

SECONDARY OUTCOMES:
characterize the peak of serum concentration (Cmax) | From pre-dose to Day70 for single dose part. From pre-dose to Day98 for multiple dose part
  evaluate the maximum observed serum concentration(Cmax) via LAE103 injection mono or LAE102 combined with LAE103 injection
characterize the time of reaching peak of serum concentration (Tmax) | From pre-dose to Day70 for single dose part. From pre-dose to Day98 for multiple dose part
  evaluate what time to reach the maximum serum concentration(Tmax)
characterize the area under the serum concentration versus time curve (AUC) | From pre-dose to Day70 for single dose part. From pre-dose to Day98 for multiple dose part
  Evaluate the area under the serum concentration versus time curve (AUC) in LAE103 mono injection or LAE102 combined with LAE103 injection
Evaluate the expression levels of Activin A in blood samples | From pre-dose to Day70 for single dose part. From pre-dose to Day98 for multiple dose part.
  The validated methodology was employed to assay serum levels of Activin A in biological samples.
Incidence of positive Anti-drug antibody(ADA) after administration | From pre-dose to Day70 for single dose part. From pre-dose to Day98 for multiple dose part.
  Test ADA status in biological sample via validated methodology

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wong, Principal Investigator — Q-Pharm Pty Ltd.
Locations (1):
- Q-Pharm Pty Ltd., Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No